CLINICAL TRIAL: NCT01879891
Title: Exercise Intensity, Metabolic Rate and Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Gary Hunter, PhD, Gary R. Hunter, PhD, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 5R01DK049779-14 (NIH)
Record Dates: First submitted 2013-06-13; First posted 2013-06-18 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Healthy Women
Keywords: Exercise Intensity; Metabolism; Insulin
MeSH Terms: conditions — Insulin Resistance

ARMS (2):
- Non-Biopsy (Other): The Non-Biopsy group will complete a VO2 maximum test, are provided food 2 days prior to assessments, exercise in the metabolic chamber, have a Resting Energy Expenditure test, complete a DEXA and have blood drawn. This group will stay overnight in the metabolic chamber and have the clamp procedure. Exercise training is exactly the same for both groups.
  Those who select the Non-Biopsy group, in lieu of the biopsy test, will complete an Activities of Daily Living (ADL) test that involves sub-maximal VO2 assessment. The participants will also be asked to where an accelerometer home for 4 consecutive days after the ADL test.
  Interventions: Other: Aerobic
- Biopsy (Other): The Biopsy group will also complete a VO2 maximum test, are provided food 2 days prior to assessments, exercise in the metabolic chamber, have a Resting Energy Expenditure test, complete a DEXA and have blood drawn. As with the Non-Biopsy group, this group will stay overnight in the metabolic chamber and have the clamp procedure. Exercise training is exactly the same for both groups. One week following the overnight metabolic chamber visit, participants in this group will undergo a muscle biopsy. This group will not complete the Activities of Daily Living (ADL) test nor will they be asked to wear an accelerometer.
  Interventions: Other: Aerobic

INTERVENTIONS:
Other: Aerobic — Exercise training will consist of bicycle ergometer riding starting at 67% of heart rate max for 20 minutes. Exercise Intensity will be progressively increased every week until 80% of heart rate max for 40 minute sessions is reached.

SUMMARY:
The primary goal is to test the hypothesis high interval exercise increases energy expenditure and Insulin sensitivity more than 2 days of rest or moderate intensity exercise cumulatively over 23 hours during and following the exercise. Secondary goals are to evaluate exercise difficulty during moderate intensity exercise and high interval exercise as well as difficulty of activities of daily living and free living physical activity following rest, moderate intensity exercise and high interval exercise.

A secondary study is designed to evaluate potential mechanism. Hypotheses are that changes in muscle lipid metabolism, mitochondrial function, fat and cellular insulin signals will be increased following the high intensity interval exercise. In addition, these changes will be related to changes in insulin sensitivity and increases in protein metabolism and muscle damage.

ELIGIBILITY:
Inclusion Criteria:

* healthy premenopausal African-American or Caucasian women ages 19 - 42

Exclusion Criteria:

* subjects cannot be smoking,
* taking medications which alter energy expenditure or fuel utilization,
* be diabetic or have a body mass index (BMI) less than 18 or more than 35.
* Also subjects cannot be pregnant or have cardiopulmonary disease.

Ages: 19 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 1995-05; Primary Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Exercise Intensity | 16 weeks
  To test the hypothesis that high interval exercise increases energy expenditure and Insulin sensitivity more than 2 days of rest or moderate intensity exercise cumulatively over 23 hours during and following the exercise

SECONDARY OUTCOMES:
Exercise Difficulty | 16 weeks
  To evaluate exercise difficulty during moderate intensity exercise and high interval exercise as well as difficulty of activities of daily living and free living physical activity following rest, moderate intensity exercise and high interval exercise

CONTACTS AND LOCATIONS:
Locations (1):
- UAB, Birmingham, Alabama, United States